CLINICAL TRIAL: NCT04189523
Title: Prospective Non-Randomized Interventional Pilot Study of the Effects of Early Administration of Ultrasound Guided Regional Anesthesia for Long Bone Fractures on Long Term Patient Opioid Usage
Brief Title: Does Early Administration of Ultrasound Guided Regional Anesthesia for Long Bone Fractures Effect Long Term Patient Opioid Usage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Robert Ehrman, Volunteer Faculty, Wayne State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 022419MP2F
Record Dates: First submitted 2019-12-02; First posted 2019-12-06 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Bone Fracture; Opioid Use; Opioid Dependence
Keywords: Ultrasound; Trauma; Bone Fracture; Opioid
MeSH Terms: conditions — Fractures, Bone; Opioid-Related Disorders; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: We will perform a small prospective non-randomized interventional pilot study to assess feasibility of a future full scale RCT to test our hypotheses. Interventional study subjects will be compared to controls enrolled simultaneously during the study period who meet the inclusion criteria and do not have documentation of one of the exclusion criteria. We will enroll subjects 2 controls to 1 intervention to ensure the ability to select controls as similar to the intervention population as possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care Pain Management (Active Comparator)
  Interventions: Other: SOC Pain Management
- Early Administration of US Guided Nerve Blocks (Experimental)
  Interventions: Procedure: Early US Guided Nerve Block Administration

INTERVENTIONS:
Other: SOC Pain Management — Study subjects will be compared to historical controls selected for same age +/- 5yrs, gender, fracture type who meet the inclusion criteria and do not have historical documentation of one of the exclusion criteria. Controls will be identified by the ICD-10 injury codes selected for use in this study. Clinical course and pain management data will be collected through the EMR only.
  Arms: Standard of Care Pain Management
Procedure: Early US Guided Nerve Block Administration — US-Guided regional anesthesia (fascia illiaca compartment block or brachial plexus block)
  Arms: Early Administration of US Guided Nerve Blocks

SUMMARY:
Administration of ultrasound guided peripheral nerve blocks is a procedural skill set that falls within the scope of Emergency Medicine practice. Extrapolating evidence from Anesthesia and Orthopedic literature (which shows decreased post-operative opioid use by surgical patients who receive regional anesthesia as part of their pre and perioperative pain management strategy) the investigators believe that early administration of regional anesthesia for long bone fractures by providers in the ED may have an as of yet unidentified positive impact on long term opioid use. If this is indeed found to be the case, early administration of regional anesthesia for extremity fractures would represent an area of focus for ED providers in the national effort by the medical community to combat opioid abuse.

DETAILED DESCRIPTION:
The investigators will perform a small prospective non-randomized interventional pilot study to assess feasibility of a future full scale RCT to test the hypotheses. Interventional study subjects will be compared to controls enrolled simultaneously during the study period who meet the inclusion criteria and do not have documentation of one of the exclusion criteria. The investigators will enroll subjects 2 controls to 1 intervention to ensure the ability to select controls as similar to the intervention population as possible. The study is powered for an alpha of 0.9 and an effect size (standardized difference) of 0.2. The total subjects needed to enroll is 36 with 18 subjects in each arm of the study. However, in an attempt to obtain controls as closely matched to our intervention group as possible 36 controls will be enrolled.

A. Subject Selection

Intervention subjects will be enrolled as a convenience sample when physicians participating in the study are available in the ED. Controls will be enrolled when no study participating physicians are available in the ED. Potential subjects will be selected for enrollment by research team members directly from the trauma bay or from the tracking board when they are identified as having a qualifying fracture. They will be screened for exclusion and inclusion criteria by the research assistants. The goal will be to enroll patients within 2 hours of arrival in the ED.

Inclusion Criteria:

* patients 18 years of age or older
* presentation to the emergency department with isolated fractures of the hip or proximal femur, mid or distal humerus, radius, or ulna
* poly-trauma patients with one of the previously listed fractures who do not meet exclusion criteria

Exclusion Criteria:

* Allergy to upivacaine/ropivicaine or other amide anesthetics
* evidence of compartment syndrome on exam by physician
* infection over injection site
* previously documented opioid abuse or dependence in the last year as documented in the EMR or self-reported by the patient
* current documented opioid prescription in the EMR
* patient is intubated or unable to provide consent
* poly-trauma patients with abdominal, thoracic or neurologic injury requiring operative intervention at the time of presentation to the ED

  3a. Consent: If the patient qualifies for study inclusion a research assistant will obtain patient written consent to: receive a nerve block placed by a trained physician participating in the study, allow for access of their medical record for purposes of data collection for the study and collect patient contact information for follow up communication related to the study after discharge. The patient will be informed that should they complete all the follow up information as part of this study they will receive a monetary incentive for participation in person at their final follow up, 30 days after the nerve block.

After patients are consented either a supraclavicular brachial plexus block or fascia iliaca nerve block (determined by site of injury) will be performed by an ultrasound trained faculty member, ultrasound fellow or resident who has undergone specific training to perform the blocks included in this study. The research team will be given a list of physicians qualified to perform the selected blocks for this study.

B. Interventions

Prior to administering a nerve block to an enrolled patient a complete neurovascular exam will be performed and documented on a paper form that will be kept in the patient's chart for review by orthopedic surgery and/or trauma surgery if needed while the patient is admitted. Any questionable exam findings will be discussed in conjunction with orthopedic surgery and/or trauma surgery prior to block administration.

1. b. Supraclavicular block Investigators will follow the techniques outlined by Gamo et al and NYSORA (New York School of Regional Anesthesia) for placement of supraclavicular blocks [9,21]. Patients will be placed in the supine position on a stretcher, with their arms by their sides and head rotated to the side opposite to that of their injury, at an angle of 45° from the midline. There will be continuous cardiac and pulse oximetry monitoring throughout the procedure. Towels may be placed under the shoulder on the side of the injection to improve neck exposure for block placement. The neck will be prepped with Chlorhexidine antiseptic and sterile technique will be utilized during block placement. Blocks will be performed under ultrasound guidance using a high frequency linear probe on a Zonare machine with a sterile probe cover. The ultrasound probe will be positioned behind the clavicle in the supraclavicular fossa and pointed inferior-medially. The subclavian artery will be identified in the short axis by its rounded shape and pulsatility. The brachial plexus in this location will be identified by its proximity to the subclavian artery as it typically lies superficial and posterior-lateral to this vessel. Once the plexus is identified a clip of the plexus will be saved and uploaded to QPath for documentation. A local skin wheal of 0.5% bupivacaine will be made with a 27-guage needle 2 cm lateral to the US probe at the site of entry for the nerve block. An 'in-plane' technique will be used for visualizing the needle for block placement. A 20 or 22-gauge non-cutting needle will be introduced from lateral to medial and placed in-line with and parallel to the probe. The needle will inserted deep between the subclavian artery and the first rib, inferior to the brachial plexus; subsequently, 2 ml to 3 ml of 0.5% Bupivacaine will be injected very carefully to avoid accidental intravascular injection. The needle will be redirected from deep to intermediate and superficial levels in order to allow maximum spread of local anesthetic around the nerve bundle. By the end of the procedure, a total of 20 ml to 25 ml of 0.5% bupivacaine local anesthetic will be injected. A second clip will be saved on the Zonare and uploaded to QPath after completing the block to demonstrate the area of anesthetic introduced. Following block application patient will receive care for their injury as determined by their EM physician while in the ED and/or their admitting physician if admitted to the hospital.
2. b. Fascia Iliaca block Investigators will follow the techniques outlined by Beaudoin et al and NYSORA for placement of Fascia Iliaca blocks [13, 22]. There will be continuous cardiac and pulse oximetry monitoring throughout the procedure. Patient will be positioned supine on a stretcher in slight trendelenberg. Blocks will be performed under ultrasound guidance using a high frequency linear probe on a Zonare machine with a sterile probe cover. The inguinal region on the corresponding side of injury will be prepped with Chlorhexidine antiseptic and sterile technique will be utilized during block placement. The US probe will be placed 1 cm distal to the inguinal ligament on the side of the injured lower extremity to identify the femoral vessels and the nerve in cross section. The nerve will be identified as an isolated hyperechoic structure approximately 1 cm lateral to the pulsatile femoral artery. A clip of the identified nerve will be saved and uploaded to QPath for documentation. A local skin wheal of 0.5% bupivacaine will be made with a 27-guage needle 2 cm lateral to the US probe at the site of entry for the nerve block. At the skin wheal site, a 20 or 22-gauge noncutting spinal needle will be introduced at a 45° angle in-plane to the US probe and 20-25 mL of 0.5% bupivacaine will injected along the nerve sheath. The needle will be directly visualized throughout the procedure to ensure there is no vascular puncture and that spread of 0.5% Bupivacaine is administered in the correct fascial plane. A second clip will be saved on the Zonare and uploaded to QPath after completing the block to demonstrate the area of anesthetic introduced. Following block application patient will receive care for their injury as determined by their EM physician while in the ED and/or their admitting physician if admitted to the hospital.
3. b. Procedure Risks The possible risks associated with placement of nerve blocks while low in incidence, include possible risk of injury to vascular or nerve structures or accidental intravascular deposition of anesthetic [8,9,13,21,22]. Additional risk with the supraclavicular block includes a slight chance for pneumothorax. By placing these nerve blocks with ultrasound guidance it significantly reduces the risk of the aforementioned complications as the needle tip location is constantly visualized on screen [8,21,22]. This including decreasing the risk for pneumothorax with the supraclavicular block as the lung pleura and needle tip can be continuously visualized by ultrasound and thus help avoid accidental puncture [8,9,21]. Additionally, investigators will utilize non-cutting spinal needles for this study as this measure has been noted in previous nerve block studies to reduce the risk of accidental venous or arterial puncture and lessens the chance of injury to the epineurium of nerve bundles [9,13,21,22]. There is always the risk of allergy to bupivacaine though this is rare. Investigators will attempt to avoid allergic reactions by patients undergoing blocks by screening for allergy to amide anesthetics (the family of drugs that Bupivacaine belongs to) at time of enrollment.

C. Subject Follow Up

1. c. First 24hrs All study patients will have a reported pain score assessed using a validated pain score tool (VAS) by the research team once prior to leaving the ED. A research assistant will obtain a patient reported pain score at 24hrs after block application. While patient is admitted their utilized opioid pain medications will be tracked in the EMR and their daily MME usage will be calculated and recorded. The investigators will evaluate patient opioid usage by calculating Morphine Milligram Equivalents using CMS guidelines for conversion.
2. c. Follow up at 1 week At 7 days after block placement patients will be contacted by phone by the research team or in person if they are still hospitalized. Assistants will ask patients to report a pain score for their injury, any new injuries requiring opioid pain medication since discharge, and current opioid usage via prescribed narcotics or illicit drug use. The patient will be asked to report a pill count of their current opioid prescription (if any). Pharmacy reported prescriptions will be pulled for each patient at 7 days after initial block placement using the "External Rx History" tab under power orders in the EMR. The investigators will evaluate patient opioid usage by calculating Morphine Milligram Equivalents using CMS guidelines for conversion. At that time subjects who received a nerve will also be asked questions regarding their satisfaction with their pain control and care after receiving the nerve blocks. Subjects who did not receive a nerve block will be asked the same questions about satisfaction with pain control and will be asked about satisfaction with their care. All subjects will be asked if they have scheduled any doctor's appointments or presented to an urgent care or emergency department for the sole purpose of obtaining care for pain control for their injury.
3. c. Final follow up at 30 days At 30 days after block placement patients will be contacted by phone for a final survey by the research team. If subjects are still hospitalized they will be assessed by a research assistant in the hospital. Assistants will ask patients to report a pain score for their injury, any new injuries requiring opioid pain medication since discharge, and current opioid usage via prescribed narcotics or illicit drug use. The patient will be asked to report a pill count of their current opioid prescription (if any). Pharmacy reported prescriptions will be pulled for each patient at 30 days after initial block placement using the "External Rx History" tab under power orders in the EMR. Investigators will evaluate patient opioid usage by calculating Morphine Milligram Equivalents using CMS guidelines for conversion. At that time subjects who received a nerve will also be asked questions regarding their satisfaction with their pain control and care after receiving the nerve blocks. Subjects who did not receive a nerve block will be asked the same questions about satisfaction with pain control and will be asked about satisfaction with their care. All subjects will be asked if they have scheduled any doctor's appointments or presented to an urgent care or emergency department for the sole purpose of obtaining care for pain control for their injury. At the time of this final follow up participating patients will receive an incentive gift card for participation. Transportation to this final follow up visit will be arranged and paid for by the research department.

D. Data Collection and Interpretation

Data on each subject will be collected by research assistants and stored in a secure, de-identified REDCap database/spreadsheet. Data points collected will include: age, sex, fracture type, history of opioid abuse or opioid prescription, history if IV drug use, type of nerve block administered, and location of block placement. At follow up points data will be collected on patient reported pain scores using the VAS scoring system. Self reported opioid use, pill counts and reported healthcare visits for pain from initial injury will be recorded and stored. Data will be collected at follow ups on patient satisfaction using surveys that have Likert scaled questions. Data will be collected directly from the EMR at previously outlined points documenting each subjects opioid prescriptions and opioid use.

A statistician from the Wayne State Research Department will be utilized for data interpretation after collection of data from subjects.

E. Study Timeline

This pilot study will be conducted over a span of 12 months. The initial 6 weeks will be utilized providing study training to the participating research assistants. This time will also be spent providing block training, skills assessments and teaching to participating physicians. The following 8 months will be spent enrolling subjects and collecting data. The remaining 2 months and 2 weeks will be used for data interpretation and creation of a manuscript for submission detailing findings from this study.

ELIGIBILITY:
Inclusion Criteria:

* patients 18 years of age or older
* presentation to the emergency department with isolated fractures of the hip or proximal femur, mid or distal humerus, radius, or ulna
* poly-trauma patients with one of the previously listed fractures who do not meet exclusion criteria

Exclusion Criteria:

* Allergy to Bupivacaine/ropivicaine or other amide anesthetics
* evidence of compartment syndrome on exam by physician
* infection over injection site
* previously documented opioid abuse or dependence in the last year as documented in the EMR or self-reported by the patient
* current documented opioid prescription in the EMR
* patient is intubated or unable to provide consent
* poly-trauma patients with abdominal, thoracic or neurologic injury requiring operative intervention at the time of presentation to the ED

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Opioids administered for pain control as measured in Morphine Milliequivalents | 24-hours following injury
  Determine if early administration of nerve blocks results in change in morphine milliequivalents (MMEs) required for pain control compared to standard care.

SECONDARY OUTCOMES:
Opioids administered for pain control as measured in Morphine Milliequivalents | 7-days following injury
  Determine if early administration of peripheral nerve blocks results in change in MMEs required for pain control compared to standard care.
Opioids administered for pain control as measured in Morphine Milliequivalents | 30-days following injury
  Determine if early administration of nerve blocks results in change in MMEs required for pain control compared to standard care.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ehrman, MD, Principal Investigator — Wayne SU
Locations (2):
- United States (2):
  - Detroit Receiving Hospital, Detroit, Michigan
  - Sinai Grace Hospital, Detroit, Michigan

REFERENCES:
- [Background] Delgado MK, Huang Y, Meisel Z, Hennessy S, Yokell M, Polsky D, Perrone J. National Variation in Opioid Prescribing and Risk of Prolonged Use for Opioid-Naive Patients Treated in the Emergency Department for Ankle Sprains. Ann Emerg Med. 2018 Oct;72(4):389-400.e1. doi: 10.1016/j.annemergmed.2018.06.003. Epub 2018 Jul 24. PMID 30054152
- [Background] Dixit V, Fathima S, Walsh SM, Seviciu A, Schwendt I, Spittler KH, Briggs D. Effectiveness of continuous versus single injection femoral nerve block for total knee arthroplasty: A double blinded, randomized trial. Knee. 2018 Aug;25(4):623-630. doi: 10.1016/j.knee.2018.04.001. Epub 2018 Apr 26. PMID 29705075
- [Background] Mohamadi A, Chan JJ, Lian J, Wright CL, Marin AM, Rodriguez EK, von Keudell A, Nazarian A. Risk Factors and Pooled Rate of Prolonged Opioid Use Following Trauma or Surgery: A Systematic Review and Meta-(Regression) Analysis. J Bone Joint Surg Am. 2018 Aug 1;100(15):1332-1340. doi: 10.2106/JBJS.17.01239. PMID 30063596
- [Background] Thong ISK, Jensen MP, Miro J, Tan G. The validity of pain intensity measures: what do the NRS, VAS, VRS, and FPS-R measure? Scand J Pain. 2018 Jan 26;18(1):99-107. doi: 10.1515/sjpain-2018-0012. PMID 29794282
- [Background] Hah JM, Bateman BT, Ratliff J, Curtin C, Sun E. Chronic Opioid Use After Surgery: Implications for Perioperative Management in the Face of the Opioid Epidemic. Anesth Analg. 2017 Nov;125(5):1733-1740. doi: 10.1213/ANE.0000000000002458. PMID 29049117
- [Background] Compton WM, Jones CM, Baldwin GT. Relationship between Nonmedical Prescription-Opioid Use and Heroin Use. N Engl J Med. 2016 Jan 14;374(2):154-63. doi: 10.1056/NEJMra1508490. No abstract available. PMID 26760086
- [Background] Ritcey B, Pageau P, Woo MY, Perry JJ. Regional Nerve Blocks For Hip and Femoral Neck Fractures in the Emergency Department: A Systematic Review. CJEM. 2016 Jan;18(1):37-47. doi: 10.1017/cem.2015.75. Epub 2015 Sep 2. PMID 26330019
- [Background] Lewis SR, Price A, Walker KJ, McGrattan K, Smith AF. Ultrasound guidance for upper and lower limb blocks. Cochrane Database Syst Rev. 2015 Sep 11;2015(9):CD006459. doi: 10.1002/14651858.CD006459.pub3. PMID 26361135
- [Background] Gamo K, Kuriyama K, Higuchi H, Uesugi A, Nakase T, Hamada M, Kawai H. Ultrasound-guided supraclavicular brachial plexus block in upper limb surgery: outcomes and patient satisfaction. Bone Joint J. 2014 Jun;96-B(6):795-9. doi: 10.1302/0301-620X.96B6.31893. PMID 24891581
- [Background] Andreae MH, Andreae DA. Regional anaesthesia to prevent chronic pain after surgery: a Cochrane systematic review and meta-analysis. Br J Anaesth. 2013 Nov;111(5):711-20. doi: 10.1093/bja/aet213. Epub 2013 Jun 28. PMID 23811426
- [Background] Beaudoin FL, Haran JP, Liebmann O. A comparison of ultrasound-guided three-in-one femoral nerve block versus parenteral opioids alone for analgesia in emergency department patients with hip fractures: a randomized controlled trial. Acad Emerg Med. 2013 Jun;20(6):584-91. doi: 10.1111/acem.12154. PMID 23758305
- [Background] Haines L, Dickman E, Ayvazyan S, Pearl M, Wu S, Rosenblum D, Likourezos A. Ultrasound-guided fascia iliaca compartment block for hip fractures in the emergency department. J Emerg Med. 2012 Oct;43(4):692-7. doi: 10.1016/j.jemermed.2012.01.050. Epub 2012 Apr 9. PMID 22494596
- [Background] Beaudoin FL, Nagdev A, Merchant RC, Becker BM. Ultrasound-guided femoral nerve blocks in elderly patients with hip fractures. Am J Emerg Med. 2010 Jan;28(1):76-81. doi: 10.1016/j.ajem.2008.09.015. PMID 20006206
- [Background] Stone MB, Price DD, Wang R. Ultrasound-guided supraclavicular block for the treatment of upper extremity fractures, dislocations, and abscesses in the ED. Am J Emerg Med. 2007 May;25(4):472-5. doi: 10.1016/j.ajem.2006.08.019. PMID 17499669
- [Background] Foss NB, Kristensen BB, Bundgaard M, Bak M, Heiring C, Virkelyst C, Hougaard S, Kehlet H. Fascia iliaca compartment blockade for acute pain control in hip fracture patients: a randomized, placebo-controlled trial. Anesthesiology. 2007 Apr;106(4):773-8. doi: 10.1097/01.anes.0000264764.56544.d2. PMID 17413915
- [Background] Fletcher AK, Rigby AS, Heyes FL. Three-in-one femoral nerve block as analgesia for fractured neck of femur in the emergency department: a randomized, controlled trial. Ann Emerg Med. 2003 Feb;41(2):227-33. doi: 10.1067/mem.2003.51. PMID 12548273
- [Background] American Academy of Orthopaedic Surgeons. 2014. Strong evidence supports regional analgesia to improve preoperative pain control in patients with hip fracture. Retrieved from: http://www.orthoguidelines.org/guideline-detail?id=1231
- [Background] T Bendinger, N Plunkett; Measurement in pain medicine, BJA Education, Volume 16, Issue 9, 1 September 2016, Pages 310-315, https://doi.org/10.1093/bjaed/mkw014
- [Background] A Feizerfan, G Sheh; Transition from acute to chronic pain, Continuing Education in Anaesthesia Critical Care & Pain, Volume 15, Issue 2, 1 April 2015, Pages 98-102, https://doi.org/10.1093/bjaceaccp/mku044
- [Background] Key Substance Use and Mental Health Indicators in the United States: Results from the 2016 National Survey on Drug Use and Health: pages 20-24. Center for Behavioral Health Statistics and Quality, US Dept Health and Human Services; 2016. https://www.samhsa.gov/data/sites/default/files/NSDUH-FFR1-2016/NSDUH-FFR1-2016.pdf